CLINICAL TRIAL: NCT06701292
Title: Precision Ablation For Pulmonary Vein Isolation: Targeting Pulmonary Vein Myocardial Sleeves With Omnipolar Mapping Technology - A Randomized Pilot Trial
Brief Title: Precision Ablation For Pulmonary Vein Isolation: Targeting Pulmonary Vein Myocardial Sleeves (PVMS) With Omnipolar Mapping Technology
Acronym: PVS-PVI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment after technological advances replaced the study procedure.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ramesh Hariharan, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-24-0150
Record Dates: First submitted 2024-11-17; First posted 2024-11-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; symptomatic paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PVS-PVI (Experimental)
  Interventions: Device: PVS-PVI targeted ablation
- WACA (Active Comparator)
  Interventions: Device: Wide area circumferential ablation (WACA)

INTERVENTIONS:
Device: PVS-PVI targeted ablation — Omnipolar technology will be used to analyze all PVs and delineate the PVMS. Once identified, PVMS will be marked and described in a clockface fashion using a lateral view of the vein.Ablation will target the PVMS using the same power and force parameters as described for the WACA procedure. Effective ablation lesions and distance between ablation spots will be represented in the same manner too. Lesions should cover at least 5 mm outside the PVMS delineation on both PVMS borders of each myocardial sleeve. PVI will be demonstrated with the same technique described in the WACA procedure.
  The PVI will be verified for each vein 10 minutes after the initial achievement of PVI.
  Arms: PVS-PVI
Device: Wide area circumferential ablation (WACA) — After generating the 3D electroanatomical map of the heart to understand where treatment needs to be applied,using a tool called radiofrequency (RF) ablation, small burns will be made around the veins to block abnormal electrical signals. Each burn is applied with up to 50 watts of power and lasts up to 10 seconds.The ablation tool will press down with a force of around 10-20 grams.The mapping system (NAVX software) shows the burns on the 3D map
  Arms: WACA

SUMMARY:
The purpose of this study is to compare procedural times and Radiofrequency (RF)applications required for Pulmonary vein myocardial sleeves targeted pulmonary vein ablation (PVS-PVI) , to compare the efficacy of PVS-PVI , to compare the safety of PVS-PVI and to assess other clinical outcomes of PVS-PVI in individuals with symptomatic paroxysmal Atrial fibrillation (AF) using Omnipolar Technology with conventional Wide area circumferential ablation (WACA).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal AF refractory to at least one Class I or Class III antiarrhythmic medication, intolerance to antiarrhythmic medications, or a preference to not trial antiarrhythmic medications
* A minimum of one documented AF episode via 12-lead ECG, Holter monitor, or loop recorder
* Capability to provide informed consent

Exclusion Criteria:

* Persistent or permanent AF
* Prior history of catheter or surgical ablation for AF or left atrial ablation for atypical flutter
* Reversible causes of AF
* Congenital heart disease
* Significant valve disease (moderate or severe mitral/aortic stenosis or regurgitation)
* Pregnancy
* Known presence of intracardiac thrombus
* Systemic oral anticoagulation therapy contraindicated, including a history of heparin-induced thrombocytopenia
* Broad vortex-like connections and no clear PVMS to be targeted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of minutes taken from Initial puncture to transseptal access | From time of Initial puncture to time of transseptal access (an average of 10 minutes)
Number of minutes taken from transseptal access to left atrium 3D map completion | From time of transseptal access to time of left atrium 3D map completion (an average of 15 minutes)
Number of minutes taken from left atrium 3D map completion to when all pulmonary veins are isolated | From time of left atrium 3D map completion to time when all pulmonary veins are isolated (an average of 30-60 minutes)
Number of minutes with catheters in the left atrium | from time catheters are inserted to time catheters are removed (an average of 45-80 minutes)
Time from initial puncture till all sheaths removed | From time of initial puncture to time when all sheaths removed (an average of 90 minutes)
Total time of radiofrequency applications in seconds | from start of radiofrequency application to end of radiofrequency applications(an average of 300-900 seconds)
Number of radiofrequency applications used | end of procedure (an average of 1.5 hours after baseline)

SECONDARY OUTCOMES:
Day and time to first recurrence of any documented atrial arrhythmias | an average of 91 days after catheter ablation
  This will be remotely monitored with the Internal loop recorder (ILR) monthly and in clinic every 3 months until the end of the follow up
Time in sinus rhythm as assessed by the percentage of time that the patient remains in sinus rhythm during the pre-established monitoring | 3 months follow up
  This will be remotely monitored with the ILR monthly and in clinic every 3 months until the end of the follow up
Time in sinus rhythm as assessed by the percentage of time that the patient remains in sinus rhythm during the pre-established monitoring | 6 months follow up
  This will be remotely monitored with the ILR monthly and in clinic every 3 months until the end of the follow up
Number of Procedure-related complications | end of study (6 months after procedure)
  Complications include Atrio-esophageal fistula, Stroke or transient ischemic attack (TIA), Pericardial effusion/cardiac tamponade, PV stenosis , Vascular access-related complications , Diaphragmatic paralysis , other severe complications or other non-severe complications 0.37%
Number of deaths | end of study (6 months after procedure)
Total radiation exposure dose | end of procedure (about 1.5 hours after start of procedure)
Number of participants that need a repeat catheter ablation procedure due to documented recurrence of symptomatic atrial arrhythmia | end of procedure till 6 months after procedure
Number of occurrences of any AF (symptomatic or asymptomatic) documented on ECG or ILR | during the first 90 days following catheter ablation.
Number of participants that visit the emergency room | end of procedure till 6 months after procedure
Number of participants that are hospitalized | end of procedure till 6 months after procedure
Number of incidences of stroke | end of procedure till 6 months after procedure
Change in quality of life as assessed by the Quality of Life (EQ-5D-5L) assessment | Baseline, 6 months after procedure
  This is a 6 item questionnaire and the first 5 questions are each is scored from 1(no problem)-5(unable to) for a maximum score of 25, higher number indicating worse outcome. The 6th question is score on likert scale from 0(worst health you can imagine)-100(best health you can imagine), higher score indicating worse outcome
Number of participants that show a need for electrical cardioversion | end of procedure till 6 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Hariharan, D, MRCP,FACC, FHRS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No